CLINICAL TRIAL: NCT05856513
Title: A Phase I Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of ZSP1273
Brief Title: Pharmacokinetics of ZSP1273 in Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ZSP1273-23-12
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Hepatic Impairment; Pharmacokinetics
MeSH Terms: interventions — ZSP1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child-Pugh A (Experimental): 8 participants with mild hepatic impairment (Child-Pugh A) will be given 600mg of ZSP1273.
  Interventions: Drug: ZSP1273
- Child-Pugh B (Experimental): 8 participants with moderate hepatic impairment (Child-Pugh B) will be given 600mg of ZSP1273.
  Interventions: Drug: ZSP1273
- Normal hepatic function (Experimental): 8 participants with normal hepatic function will be given 600mg of ZSP1273.
  Interventions: Drug: ZSP1273

INTERVENTIONS:
Drug: ZSP1273 — Participants receive ZSP1273 orally.
  Arms: Child-Pugh A
Drug: ZSP1273 — Participants receive ZSP1273 orally.
  Arms: Child-Pugh B
Drug: ZSP1273 — Participants receive ZSP1273 orally.
  Arms: Normal hepatic function

SUMMARY:
This study will assess the effect of hepatic impairment on the pharmacokinetics (PK), safety and tolerability of ZSP1273.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 to ≤ 68 years, at the time of signing the informed consent.
2. BMI ≥ 18 kg/m2 up to ≤ 32 kg/m2.
3. Participants (including partners) must use reliable methods of contraception during the study and until 3 months following the last dose of investigational product.
4. Signature of a dated Informed Consent Form (ICF) indicating that the participates has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.

   Participants with hepatic impairment only:
5. Supporting documents confirming that the participant has liver cirrhosis with hepatic impairment must be available.
6. Unless otherwise stated, participants must have been on stable doses and regimens of the concomitant medication for at least 4 weeks before screening, or treatment-naïve participants

Exclusion Criteria:

1. Participants with an allergic disposition (multiple drug and food allergies) or who, as determined by the investigator, are likely to be allergic to the investigational drug product or any component of the investigational drug product.
2. QTcF (male) > 470ms，QTcF (female) > 480ms
3. Participants with serious infections, trauma, gastrointestinal surgery or other major surgical procedures within 4 weeks
4. Participants who donated blood or bleeding profusely (> 400 mL) in the 3 months.
5. Pregnant or lactating women, or women of childbearing age with a positive pregnancy test
6. Smoking averaged more than 10 cigarettes per day in the 3 months prior to screening

   Participants with Normal Hepatic Function Only:
7. Any history of hepatic impairment, or potential presence of liver function impairment by physical examination and laboratory examination at screening.

   Participants with Hepatic Impairment Only:
8. Any history of clinically serious illness or disease or condition except for primary liver disease that the investigator believes may affect the results of the trial, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary, respiratoryor hematological, immune, psychiatric, and metabolic disorders.
9. Participants with drug-induced liver injury; history of liver transplantation; cirrhosis in combination with the following complications: including but not limited to liver failure, hepatic encephalopathy, hepatocellular carcinoma, esophageal bleeding from ruptured fundic varices

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 to Day 6
  The Cmax of a single dose of ZSP1273 in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Area under the concentration-time curve from time zero to infinity (AUCinf) | Day 1 to Day 6
  The AUCinf of a single dose of ZSP1273 in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.
Area under the concentration-time curve from time zero to last time of quantifiable concentration (AUClast) | Day 1 to Day 6
  The AUClast of a single dose of ZSP1273 in participants with impaired hepatic function and controls with normal hepatic function will be evaluated and compared.

SECONDARY OUTCOMES:
Number of participants with drug-related adverse events as assessed by CTCAE v5.0 | Day 1 to Day12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li C, Li H, Mai J, Zhang H, Wu M, Ding Y, Huang J. Single-Dose Tolerability and Pharmacokinetics of Onradivir in Chinese Patients with Hepatic Impairment and Healthy Matched Controls. J Clin Pharmacol. 2025 Feb;65(2):226-232. doi: 10.1002/jcph.6134. Epub 2024 Sep 17. PMID 39287964